CLINICAL TRIAL: NCT04542733
Title: The Efficacy of Everolimus With Reduced-dose Tacrolimus Versus Reduced-dose Tacrolimus and Leflunomide in Treatment of BK Virus Infection in Kidney Transplantation Recipient
Acronym: ELF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Suwasin Udomkarnjananun, Principle investigator, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUKT02/63
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant Infection; BK Virus Infection
Keywords: Kidney Transplantation; mTOR inhibitor; Leflunomide; BK virus
MeSH Terms: interventions — Everolimus; Leflunomide

STUDY DESIGN:
Intervention Model Description: All patients met inclusion criteria will be randomized after BK VL not respond to mycophenolic acid and tacrolimus reduction as a run-in phase for 1 month. The intervention arms include everolimus + reduced dose tacrolimus and leflunomide + reduced dose tacrolimus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mTORi with reduced-dose tacrolimus (Active Comparator): Patient will received everolimus with target trough concentration of 3-6 ng/mL and tacrolimus with target trough concentration of 2-4 ng/mL. Duration for this regimen would be at least 3 months.
  Interventions: Drug: Everolimus
- reduced-dose tacrolimus and Leflunomide (Active Comparator): Patient will receive tacrolimus with target concentration of 3-6 ng/mL with leflunomide 100 mg/day loading dose for 5 days, followed by 40 mg/day thereafter. Duration for this regimen would be at least 3 months.
  Interventions: Drug: reduced dose tacrolimus and Leflunomide

INTERVENTIONS:
Drug: Everolimus — Everolimus will be given with tacrolimus.
  Arms: mTORi with reduced-dose tacrolimus
Drug: reduced dose tacrolimus and Leflunomide — Reduced dose tacrolimus will be given with leflunomide
  Arms: reduced-dose tacrolimus and Leflunomide

SUMMARY:
BK virus infection is one of the causes of renal allograft loss in the current era. Reduction of immunsuppression is the only intervention that prooved to be effective in treating of BK virus in kidney transplant recipient. However, there are evidences from retrospective and prospective studies showed that leflunomide and mTOR inhibitor such as everolimus or sirolimus have positive outcomes in treatment of BK virus in kidney tranplant recipient. The investigators conduct the RCT to compare the efficacy of leflunomide and mTOR inhibitor everolimus, in treatment of BK virus infected patients who do not respond to immunosuppression reduction.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients at King Chulalongkorn Memorial Hospital
* age >= 18 years
* persistent BK viremia >1000 copies/mL at least 2 times in 3 weeks or single time > 10000 copies/mL

Exclusion Criteria:

* BK VL >10^5 log
* Previous BKVAN treatment
* Drug hypersensitivity to mTORi or leflunomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Plasma BK viral load change | 3 months
  3-month plasma BK viral load change from randomization

SECONDARY OUTCOMES:
Plasma BK viral load clearance rate | 1, 3, 6 months
  Percentage of patients who have negative plasma BK virus at specific time point after randomization
Acute rejection rate | 6 months
Glomerular filtration rate (GFR) change | 3, 6 months
  GFR change at specific timepoint after randomization
Chronicity score in kidney allograft | 6 months
  Banff's criteria for allograft biopsy tissue, focus on ci and ct scores ranging from 0 (no chronicity lesion) to 3 (severe chronicity lesion)
6-month plasma BK VL | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suwasin Udomkarnjananun, MD, MSc, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand